CLINICAL TRIAL: NCT00061815
Title: A Phase 3 Randomized Multicenter Study of Cetuximab, Oxaliplatin, 5-Fluorouracil, and Leucovorin vs. Oxaliplatin, 5-Fluorouracil, and Leucovorin in Subjects With Previously Treated Metastatic, EGFR-Positive Colorectal Carcinoma
Brief Title: Study of Cetuximab, Oxaliplatin, 5-FU/LV Versus Oxaliplatin, 5-FU/LV in Patients With Previously Treated Metastatic, EGFR-Positive Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Chief Medical Officer, ImClone LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA225-014; NCT00065520 (obsolete NCT alias)
Record Dates: First submitted 2003-06-04; First posted 2003-06-06 (Estimated); Last update posted 2010-04-12 (Estimated); Status verified 2010-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cetuximab+FOLFOX4 (Experimental): * Day 1 - cetuximab loading dose of 400 mg/m2 IV, infused over 2 hours; oxaliplatin (85 mg/m2) simultaneously with leucovorin (200 mg/m2), followed by 5-FU 400 mg/m2 IV bolus followed by 5-FU 600 mg/m2 as a 22-hour continuous infusion
  * Day 2 - leucovorin 200 mg/m2 followed by 5-FU 400 mg/m2 IV bolus followed by another dose of 5-FU 600 mg/m2 as a 22-hour continuous infusion
  * Day 8 - cetuximab maintenance dose of 250 mg/m2 IV infused over 60 minutes
  Interventions: Biological: cetuximab; Drug: oxaliplatin; Drug: leucovorin; Drug: 5-fluorouracil
- FOLFOX4. (Active Comparator): * Day 1 - oxaliplatin (85 mg/m2) simultaneously with leucovorin (200 mg/m2), followed by 5-FU 400 mg/m2 IV bolus followed by 5-FU 600 mg/m2 as a 22-hour continuous infusion.
  * Day 2 - leucovorin 200 mg/m2 followed by 5-FU 400 mg/m2 IV bolus followed by another dose of 5-FU 600 mg/m2 as a 22-hour continuous infusion.
  Interventions: Drug: oxaliplatin; Drug: leucovorin; Drug: 5-fluorouracil

INTERVENTIONS:
Biological: cetuximab — 400 mg/m2 IV
  Other Names: Erbitux™
  Arms: Cetuximab+FOLFOX4
Drug: oxaliplatin — 85 mg/m2 IV
  Other Names: Eloxatin®
Drug: leucovorin — 200 mg/m2 IV
  Other Names: Wellcovorin®
Drug: 5-fluorouracil — 400 mg/m2 IV
  Other Names: 5-FU
Drug: 5-fluorouracil — 600 mg/m2 IV
  Other Names: 5-FU
Biological: cetuximab — 250 mg/m2 IV
  Other Names: Erbitux™
  Arms: Cetuximab+FOLFOX4

SUMMARY:
The purpose of this study is to compare overall survival in patients with previously-treated metastatic, epidermal growth factor receptor (EGFR)-positive colorectal cancer treated with oxaliplatin, 5-fluorouracil and leucovorin (FOLFOX4) and cetuximab with FOLFOX4 alone.

ELIGIBILITY:
Inclusion Criteria:

* Documented colorectal cancer which is EGFR-positive and is metastatic.
* Prior irinotecan, alone or in combination, as first-line treatment of metastatic disease.

Exclusion Criteria:

* A serious uncontrolled medical disorder that, in the opinion of the Investigator, would impair the ability of the subject to receive protocol therapy.
* Known dihydropyrimidine dehydrogenase (DPD) deficiency.
* Known metastases in the central nervous system.
* Symptomatic sensory or peripheral neuropathy.
* More than one prior chemotherapy regimen for the treatment of metastatic colorectal cancer.
* Prior oxaliplatin therapy.
* Prior cetuximab or other therapy which targets the EGF pathway.
* Prior chimerized or murine monoclonal antibody therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2003-03; Primary Completion 2004-12 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Compare overall survival in subjects with previously-treated metastatic, epidermal growth factor receptor (EGFR)-positive colorectal cancer treated with oxaliplatin, 5-FU, and LV (FOLFOX4) and cetuximab with FOLFOX4 alone. | Every six weeks

SECONDARY OUTCOMES:
Compare the response rates between the two treatment arms. | Every six weeks
Compare progression-free survival between the two treatment arms. | Every six weeks
Duration of response within each treatment arm. | Every six weeks
Time to response within each treatment arm. | Every six weeks
Compare the safety profiles between the two treatment arms. | Every six weeks
Compare the quality of life (QOL)between the two treatment arms. | Every six weeks
Conduct an economic assessment comparing healthcare resource utilization between the two treatment arms. | Every six weeks

CONTACTS AND LOCATIONS:
Overall Officials: E-mail: ClinicalTrials@ ImClone.com, Study Chair — Eli Lilly and Company
Locations (39):
- United States (39):
  - ImClone Investigational Site, Little Rock, Arkansas
  - ImClone Investigational Site, Springdale, Arkansas
  - ImClone Investigational Site, Fountain Valley, California
  - ImClone Investigational Site, Gilroy, California
  - ImClone Investigational Site, Greenbrae, California
  - ImClone Investigational Site, Orange, California
  - ImClone Investigational Site, Pomona, California
  - ImClone Investigational Site, San Diego, California
  - ImClone Investigational Site, Vista, California
  - ImClone Investigational Site, Hartford, Connecticut
  - ImClone Investigational Site, Norwalk, Connecticut
  - ImClone Investigational Site, Stamford, Connecticut
  - ImClone Investigational Site, Waterbury, Connecticut
  - ImClone Investigational Site, Boynton Beach, Florida
  - ImClone Investigational Site, Jacksonville, Florida
  - ImClone Investigational Site, Leesburg, Florida
  - ImClone Investigational Site, Orlando, Florida
  - ImClone Investigational Site, Tampa, Florida
  - ImClone Investigational Site, Atlanta, Georgia
  - ImClone Investigational Site, Macon, Georgia
  - ImClone Investigational Site, Louisville, Kentucky
  - ImClone Investigational Site, Baton Rouge, Louisiana
  - ImClone Investigational Site, Baltimore, Maryland
  - ImClone Investigational Site, Clinton, Maryland
  - ImClone Investigational Site, Saint Joseph, Michigan
  - ImClone Investigational Site, Kansas City, Missouri
  - ImClone Investigational Site, Rolla, Missouri
  - ImClone Investigational Site, Hackensack, New Jersey
  - ImClone Investigational Site, Armonk, New York
  - ImClone Investigational Site, Brooklyn, New York
  - ImClone Investigational Site, East Setauket, New York
  - ImClone Investigational Site, Winston-Salem, North Carolina
  - ImClone Investigational Site, Bismarck, North Dakota
  - ImClone Investigational Site, Philadelphia, Pennsylvania
  - ImClone Investigational Site, Charleston, South Carolina
  - ImClone Investigational Site, Knoxville, Tennessee
  - ImClone Investigational Site, Nashville, Tennessee
  - ImClone Investigational Site, Ogden, Utah
  - ImClone Investigational Site, Richmond, Virginia